CLINICAL TRIAL: NCT02278432
Title: Evaluation of the Prophylactic Use of Omeprazole in Patients Admitted to the State Hospital of Américo Brasiliense
Status: Completed | Type: Observational
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Collaborators: Hospital Estadual Américo Brasiliense (Unknown); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Samir Antonio Rodrigues Abjaude, Master's degree student, Universidade Estadual Paulista Júlio de Mesquita Filho
Other Study IDs: 28217914.6.0000.5426
Record Dates: First submitted 2014-10-28; First posted 2014-10-30 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Omeprazole
Keywords: risk assessment; pharmacovigilance; pharmacoepidemiology; drug toxicity; adverse drug reaction reporting system; omeprazole
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Introduction. The prevalence of the use of drugs that act on the gastric system has increased in the population. Omeprazole is an inhibitor of the protons pump and has a widespread use, mainly as a prophylactic to prevent reflux esophagitis, gastric pathological hypersecretory conditions, prevention of recurrence of gastric or duodenal ulcers, gastric mucosal protection against damage caused by nonsteroidal anti-inflammatory drugs and during Zollinger-Ellison syndrome. However, omeprazole is associated with several adverse events due to abusive use or irrational prescribing, in disagreement with the indication, which may cause the ineffectiveness of the drug and decreased patient safety. Objectives. To assess the risk (occurrence of adverse events) and the benefit (effectiveness) of the prophylactic use of omeprazole in hospitalized patients and to know the reasons for the prophylactic use (indicated use or not approved). Patients and Methods. A observational and cross pharmacoepidemiological study will be performed from June to November 2014, in the General State tertiary referral Américo Brasiliense Hospital. Hospitalized patients will be separated into three groups: those who make indicated and approved prophylactic use of omeprazole (exposed group 1), those who make not indicated and not approved prophylactic use (exposed group 2), and those who do not use the omeprazole (non-exposed group). Patients who do not make prophylactic use of omeprazole will be excluded. Patients will have their pharmacotherapy monitored and data will be collected daily using an investigation guide of the first day of admission and will be included in group 1 or 2, from the first use of omeprazole to discontinuation (washout period of seven half-lives or higher). National Coordinating Council for Medication Error Reporting and Prevention (NCCMERP) algorithm will be used for causality analysis is used. Data will be tabulated according to the presence or absence of effectiveness and the presence or absence adverse events in the three groups. The odds ratio of adverse events and effectiveness of indicated and approve or not indicated and not approved prophylactic use of omeprazole will be calculated. Expected results. It is intended to know the odds ratio of adverse events in the prophylactic use of omeprazole with or without indication or use approval, and the potential indications, dosage and unapproved methods of prophylactic use in omeprazole label.

ELIGIBILITY:
Inclusion Criteria: patients in use of omeprazole prophylactic (off label or indicated use) who will be admitted at the hospital under study,

Exclusion Criteria: Patients transferred from another hospital or ward; those with prescheduled surgery; those unable to communicate (intubated, in isolation, or mentally disoriented); and those with a hospital stay ≤24 hours.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized patients will be separated into three groups: those who make indicated and approved prophylactic use of omeprazole (exposed group 1), those who make not indicated and not approved prophylactic use (exposed group 2), and those who do not use the omeprazole (non-exposed group). Patients who do not make prophylactic use of omeprazole will be excluded. Patients will have their pharmacotherapy monitored and data will be collected daily using an investigation guide of the first day of admission and will be included in group 1 or 2, from the first use of omeprazole to discontinuation (washout period of seven half-lives or higher).
Sampling Method: Non-Probability Sample
Enrollment: 427 (Actual)
Dates: Start 2014-06; Primary Completion 2014-11 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Assessment magnesium serum level | at least one day
  Level magnesium serum will be considered normal when ranged among 1.9 to 2.5 mg/dL.
Assessment of creatinine serum level | at least one day
  Creatinine serum level will be considered normal when ranged among 0,5 a1,2 mg/dL.
Assessment of urea serum level | at least one day
  Urea serum level will be considered normal when ranged among 15 a 45 mg/dL

SECONDARY OUTCOMES:
Assessment of omeprazole effectiveness and adverse drug reaction | at least one day
  Effectiveness and safety of omeprazole are going to be performed by patient report and analysis of medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia C Mastroianni, PHD, Study Chair — School of Pharmaceutical Sciences- Unesp; Tales R De Nadai, PhD, Study Chair — Hospital Estadual de Américo Brasiliense

REFERENCES:
- [Background] Varallo FR, Capucho HC, Silva Planeta Cd, Carvalho Mastroianni Pd. Possible adverse drug events leading to hospital admission in a Brazilian teaching hospital. Clinics (Sao Paulo). 2014 Mar;69(3):163-7. doi: 10.6061/clinics/2014(03)03. PMID 24626940
- [Background] Talley NJ. Risks of proton-pump inhibitors: what every doctor should know. Med J Aust. 2009 Feb 2;190(3):109-10. doi: 10.5694/j.1326-5377.2009.tb02305.x. No abstract available. PMID 19203303
- [Background] Faulhaber GA, Ascoli BM, Lubini A, Mossmann M, Rossi G, Geib G, Furlanetto TW. Serum magnesium and proton-pump inhibitors use: a cross-sectional study. Rev Assoc Med Bras (1992). 2013 May-Jun;59(3):276-9. doi: 10.1016/j.ramb.2012.12.007. Epub 2013 May 13. PMID 23680271
- [Background] Ameijeiras AH, Gonzalez BC, Zuniga VL. [A survey of gastroprotective drugs: prescription-indication in hospitalized patients]. Gac Sanit. 2007 Sep-Oct;21(5):412-5. doi: 10.1157/13110449. Spanish. PMID 17916308
- [Derived] Varallo FR, de Nadai TR, de Oliveira ARA, Mastroianni PC. Potential Adverse Drug Events and Nephrotoxicity Related to Prophylaxis With Omeprazole for Digestive Disorders: A Prospective Cohort Study. Clin Ther. 2018 Jun;40(6):973-982. doi: 10.1016/j.clinthera.2018.04.013. PMID 29759903